CLINICAL TRIAL: NCT04883658
Title: An Open Label, Randomized, Single Dose, 2-sequence, 4-period, Cross-over Clinical Trial to Evaluate the Pharmacokinetics and Tolerability of CKD-348(2) With Coadministration of CKD-828, D097 and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of CKD-348(2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A86_09BE2108
Record Dates: First submitted 2021-04-29; First posted 2021-05-12 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Period 2: CKD-348(2) - A single oral dose of 1 tablet under fasting condition
  Period 3: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Period 4: CKD-348(2) - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-348(2); Drug: CKD-828, D097, D337
- Sequence 2 (Experimental): Period 1: CKD-348(2) - A single oral dose of 1 tablet under fasting condition
  Period 2: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Period 3: CKD-348(2) - A single oral dose of 1 tablet under fasting condition
  Period 4: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Interventions: Drug: CKD-348(2); Drug: CKD-828, D097, D337

INTERVENTIONS:
Drug: CKD-348(2) — QD, PO
Drug: CKD-828, D097, D337 — QD, PO

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and Tolerability of CKD-348(2)

DETAILED DESCRIPTION:
An open label, randomized, single dose, 2-sequence, 4-period, cross-over clinical trial to evaluate the pharmacokinetics and tolerability of CKD-348(2) with coadministration of CKD-828, D097 and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥50kg (man) or 45kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who meet the blood pressure criteria during screening tests:

   * Systolic Blood Pressure: 90 to 139 mmHg
   * Diastolic Blood Pressure: 60 to 89 mmHg
4. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
5. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
6. Those who agree to contraception during the participation of clinical trial.
7. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
2. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month before the first administration of investigational products.
3. Those who donated whole blood or apheresis within 8 weeks or 4 weeks respectfully, or received blood transfusion within a month.
4. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
5. Those who exceed an alcohol and cigarette consumption than below criteria

   * Alcohol: Man_21 glasses/week, Woman_14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL)
   * Smoking: 20 cigarettes/day
6. Those who have any history of diabetic mellitus, nephropathy, biliary obstruction, shock, angioedema, cardiac insufficiency, dihydropyridine sensitivity, unstable angina, hypothyroidism.
7. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
8. Those who are deemed insufficient to participate in this clinical study by investigators.
9. Woman who are pregnant or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-348(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of CKD-348(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of CKD-348(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCinf: Area under the concentration-time curve from zero up to ∞
Tmax of CKD-348(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Tmax: Time to maximum plasma concentration
AUCt/AUCinf of CKD-348(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCt/AUCinf
T1/2 of CKD-348(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  T1/2: Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Yook-Hwan Noh, M.D., PhD., Principal Investigator — Hplus YangJi Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea